CLINICAL TRIAL: NCT02630784
Title: Efficacy and Safety of Non-invasive Ventilation by Calibrated Leak in the Treatment of Respiratory Acidosis in ICU
Acronym: VNI Versus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollement
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-A00844-43
Record Dates: First submitted 2015-09-10; First posted 2015-12-15 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Respiratory Acidosis in ICU Patients
Keywords: Non-invasive ventilation; NIV ventilator; Exhalation by a calibrated leak; ICU ventilator; Respiratory acidosis; ICU
MeSH Terms: conditions — Acidosis, Respiratory | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Homecare ventilator (Experimental): NIV with a dedicated ventilator for homecare, functioning with a turbine and with vented mask (exhalation by a calibrated leak)
  Interventions: Procedure: Non-Invasive Ventilation with Homecare ventilator
- ICU ventilator (Active Comparator): NIV with a dedicated ICU ventilator, functioning with non-vented masks and an exhalation valve.
  Interventions: Procedure: Non-Invasive Ventilation with ICU ventilator

INTERVENTIONS:
Procedure: Non-Invasive Ventilation with Homecare ventilator
  Arms: Homecare ventilator
Procedure: Non-Invasive Ventilation with ICU ventilator
  Arms: ICU ventilator

SUMMARY:
VNI Versus is a clinical, prospective, randomized, cross over study, aiming to compare two mechanical ventilators during non-invasive ventilation for patient suffering from respiratory acidosis.

This study will compare a dedicated ventilator for Non Invasive Ventilation (NIV) functioning with a turbine and with vented mask (exhalation by a calibrated leak) and a dedicated ventilator for Intensive Care Unit (ICU), functioning with non-vented masks and an exhalation valve.

Patient will be randomized before the first NIV session lasting 2 hours. After a two hours wash-out, a second NIV treatment will be delivered with the other ventilator for duration of 2 hours.

Arterial blood samples will be collected at the beginning and the end of each session of NIV. A transcutaneous captor of dioxide carbon pressure (PCO2) will also be used for patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Dioxide carbon arterial pressure > 60 mmHg
* Blood acidity (pH) <7.36

Exclusion Criteria:-Patient age under 18

* Pregnant woman
* Cognitive disorder (other than the one induced by hypercapnia)
* Acute intoxication with morphine or benzodiazepines
* Patient already equipped prior to admission with a home NIV or Continuous Positive Airway Pressure (CPAP) device
* All contraindications to NIV already described in the French Consensus Conference on NIV, from 2006.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2018-05-05 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Carbon dioxide arterial pressure (PaCO2) | After 2 hours of NIV
  Absolute decrease in carbon dioxide arterial pressure (PaCO2) after 2 hours of ventilation

SECONDARY OUTCOMES:
Arterial blood acidity (pH) after 2 hours of NIV | after 2 hours of NIV
  Correction of arterial blood acidity (pH) after 2 hours of NIV
Transcutaneous PCO2 | 6 hours
  Kinetic of the PaCO2 correction, monitored via transcutaneous PCO2 captor.
Börg dyspnea scale | 6 hours
RASS score | 6 hours
Nurse satisfaction survey | 6 hours
Patient satisfaction survey | 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Michallon, Grenoble, France

REFERENCES:
- [Background] Akada S, Takeda S, Yoshida Y, Nakazato K, Mori M, Hongo T, Tanaka K, Sakamoto A. The efficacy of dexmedetomidine in patients with noninvasive ventilation: a preliminary study. Anesth Analg. 2008 Jul;107(1):167-70. doi: 10.1213/ane.0b013e3181732dc2. PMID 18635484
- [Background] Carteaux G, Lyazidi A, Cordoba-Izquierdo A, Vignaux L, Jolliet P, Thille AW, Richard JM, Brochard L. Patient-ventilator asynchrony during noninvasive ventilation: a bench and clinical study. Chest. 2012 Aug;142(2):367-376. doi: 10.1378/chest.11-2279. PMID 22406958
- [Background] Chiumello D, Chevallard G, Gregoretti C. Non-invasive ventilation in postoperative patients: a systematic review. Intensive Care Med. 2011 Jun;37(6):918-29. doi: 10.1007/s00134-011-2210-8. Epub 2011 Mar 18. PMID 21424246
- [Background] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735
- [Background] Girault C, Bubenheim M, Abroug F, Diehl JL, Elatrous S, Beuret P, Richecoeur J, L'Her E, Hilbert G, Capellier G, Rabbat A, Besbes M, Guerin C, Guiot P, Benichou J, Bonmarchand G; VENISE Trial Group. Noninvasive ventilation and weaning in patients with chronic hypercapnic respiratory failure: a randomized multicenter trial. Am J Respir Crit Care Med. 2011 Sep 15;184(6):672-9. doi: 10.1164/rccm.201101-0035OC. PMID 21680944
- [Background] Janssens JP, Howarth-Frey C, Chevrolet JC, Abajo B, Rochat T. Transcutaneous PCO2 to monitor noninvasive mechanical ventilation in adults: assessment of a new transcutaneous PCO2 device. Chest. 1998 Mar;113(3):768-73. doi: 10.1378/chest.113.3.768. PMID 9515855
- [Background] Peter JV, Moran JL, Phillips-Hughes J, Graham P, Bersten AD. Effect of non-invasive positive pressure ventilation (NIPPV) on mortality in patients with acute cardiogenic pulmonary oedema: a meta-analysis. Lancet. 2006 Apr 8;367(9517):1155-63. doi: 10.1016/S0140-6736(06)68506-1. PMID 16616558